CLINICAL TRIAL: NCT04961827
Title: Eat Well After Cancer: a Randomized Controlled Trial of a Self-efficacy Based Dietary Intervention Among Chinese Cancer Survivors
Brief Title: A Self-efficacy Based Dietary Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a lack of manpower
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW20-622
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Self-efficacy based images (Experimental): Intervention group with self-efficacy based images sent through instant messaging biweekly for 6 times.
  Interventions: Behavioral: Self-efficacy based images through instant messaging
- Active control: knowledge based images (Active Comparator): Active control group with knowledge based images sent through instant messaging biweekly for 6 times.
  Interventions: Behavioral: Knowledge based images through instant messaging

INTERVENTIONS:
Behavioral: Self-efficacy based images through instant messaging — A total of 6 images will be sent to participants via instant messaging. Images will utilize concepts in the Theory of self-efficacy to increase dietary self-efficacy among participants and hence improve dietary quality beyond that of conventional nutrition counseling.
  Arms: Intervention: Self-efficacy based images
Behavioral: Knowledge based images through instant messaging — A total of 6 images will be sent to participants via instant messaging. Images will consist of information covered in nutrition counseling sessions, such as those related to serving sizes.
  Arms: Active control: knowledge based images

SUMMARY:
To develop and test the effectiveness of a dietary intervention aiming to enhance self-efficacy through sending images through instant messaging.

DETAILED DESCRIPTION:
Healthy eating is linked to improved survival and quality of life among cancer survivors. However, previous studies showed that most cancer survivors were not adhering to dietary recommendations despite having made changes post-diagnosis.

Conventional nutrition counseling interventions are often used in this population. However, they are labor and cost intensive and involved multiple sessions with participants. Written materials have often been used to facilitate improvements of dietary quality beyond nutrition counseling sessions but are outdated. Therefore, we propose to develop and test the effectiveness of a dietary intervention aiming to enhance self-efficacy through sending images through instant messaging. Methods to increase self-efficacy include performance accomplishment, persuasion, modelling and peer-modelling.

A prospective, randomized controlled trial design will be used to test the effectiveness of the intervention. A total of 168 adult Chinese cancer survivors, diagnosed with non-metastatic cancer (Stages 0-III), and have completed all active treatments, including surgery and adjuvant treatments such as chemotherapy and radiation therapy will be recruited.

Participants will be randomly assigned into one of two groups at a 1:1 ratio, using computer-generated block randomization sequences. The first group will be an active control group. Participants in this group will receive knowledge-based dietary information through an instant messaging applications biweekly for 6 times. The second group will be the intervention group. Participants will receive biweekly self-efficacy enhancing materials for 6 times. Materials will provide information about behavior-health link, provide information on consequences, provide instruction, and provide opportunities for social comparison. For example, the materials will provide recipe ideas and meal planning samples from fellow cancer survivors. All materials will be developed by a registered dietitian and will be consistent with published dietary guidelines for cancer survivors.

Participants will have follow-up appointments at 3 months. Their dietary quality and skin carotenoid status will be monitored. It is hypothesized that dietary quality will be better and skin carotenoid status will be higher for participants in the intervention group compared to participants in the active control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Diagnosed with cancer, non-metastatic (Stages 0-III)
* Ability to read Chinese and speak Cantonese or Putonghua/Mandarin
* Completed all active treatments, including surgery and adjuvant treatments such as chemotherapy and radiation therapy
* Attending clinic with nutrition counseling at study site

Exclusion Criteria:

* Ethnicity other than Chinese
* Diagnosed with mental, hearing, speech, or cognitive disabilities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in mean dietary quality | Baseline and 3 months
  Servings of fruit and vegetables per day, number of red meat servings per week and ratio of whole to refined grains measured by a 3-day dietary record self-completed by participants before baseline and 3-months follow-up
Changes from baseline in mean skin carotenoid reading | Baseline and 3 months
  Skin carotenoid status reading measured by a reflective spectroscopy machine

OTHER OUTCOMES:
Changes from baseline in mean self-efficacy score | Baseline and 3 months
  Dietary related self-efficacy measured by a 15-item scale (DIET-SE), consisted of 10 scenario based questions and 5 general questions.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lam, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- JCICC, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No